CLINICAL TRIAL: NCT03283605
Title: Phase I/II of Durvalumab (MEDI4736) + Tremelimumab + Stereotactic Body Radiotherapy for Metastatic Head and Neck Carcinoma
Brief Title: Immunotherapy and SBRT for Metastatic Head and Neck Carcinomas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12361
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Metastatic Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Single group assignment
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + tremelimumab and SBRT (Experimental): All subjects will receive durvalumab (1500 mg IV q4week) and tremelimumab (75mg q4week) for 4 doses, followed by durvalumab alone (1500 mg IV q4week) until disease progression, unacceptable toxicity or patient withdrawal. SBRT will be administered between cycle 2 and 3 of durvalumab and tremelimumab. All SBRT will be completed within a 3-week period.
  Interventions: Radiation: SBRT; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Radiation: SBRT — SBRT to 2-5 oligometastases will be administered between Cycle 2 and 3 of durvalumab and tremelimumab. All SBRT will be completed within a 3-week period.
Drug: Durvalumab — Durvalumab (1500 mg IV q4weeks) for 4 cycles in combination with tremelimumab. Then, durvalumab alone until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or other discontinuation criteria met.
Drug: Tremelimumab — Tremelimumab (75mg IV q4weeks) for 4 cycles in combination with Durvalumab.

SUMMARY:
Immunotherapy targeting the PD-1/PD-L1 pathway had previously been shown to be efficacious in the treatment of patients with metastatic head and neck squamous cell carcinomas. Stereotactic Body Radiotherapy (SBRT) to metastatic lesions causes localized cancer cell killing and the release of cancer cell debris, which could stimulate the immune system in the presence of immunotherapy. The purpose of this study is to assess the tolerability and efficacy of combining Durvalumab (MEDI4736), Tremelimumab and SBRT in controlling cancer progression. SBRT will be administered to patients while they are receiving Durvalumab and Tremelimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) confirmed diagnosis HNSCC at a metastatic site. This includes histologic variants of SCC such as spindle cell carcinoma, poorly differentiated keratin-positive carcinoma, and lymphoepithelioma. The pathology can come from the most accessible site and does not need to be from the time of diagnosis.
2. ≥2 locoregional and/or extracranial metastatic lesions (no brain metastases) that are treatable by SBRT. Lesions that are not measurable per RECIST v1.1 must show progression on 2 consecutive imaging studies with a minimum increase of 1 mm, and must be a mimimum size of 5 mm at time of enrollment. .
3. ≤ 4 prior treatment lines with systemic therapy
4. ≥2 measurable disease (RECIST) consisting of extracranial metastatic lesions (no brain metastasis) that are treatable by SBRT.
5. ≤ 10 metastatic lesions
6. Life expectancy > 24 weeks
7. Evaluation by a radiation oncologist within 45 days prior to study registration
8. Evaluation by a medical oncologist within 45 days prior to study registration
9. Body weight >30kg
10. The following imaging workup to document metastases within 45 days prior to study registration:

    * CT scans of the chest, abdomen and pelvis OR whole body PET/CT
11. ≥ 18 years of age at time of study entry
12. Up to 4 prior treatment lines with systemic therapy are allowed
13. Eastern Cooperative Oncology Group/World Health Organisation (ECOG/WHO) performance status score of ≤ 1
14. Patients with locoregional recurrence(s) can be included only if they have evidence of distant metastasis; patients with locoregional recurrences which are symptomatic and/or potentially affect quality of life may undergo palliative radiation therapy to this region prior to enrollment on the protocol at the discretion of the treating physician. However, a minimum of 6 weeks must elapse before receiving protocol treatment.
15. Adequate normal organ and marrow function as defined below:

    * Haemoglobin ≥ 9.0 g/dL
    * Absolute neutrophil count (ANC ≥ 1.5 (or 1.0) x (> 1500 per mm3)
    * Platelet count ≥ 100 (or 75) x 109/L (>75,000 per mm3)
    * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
    * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (calculated by study site staff)
16. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
17. Patient is willing and able to give written informed consent, prior to performing any protocol-related procedures, including screening evaluations.
18. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
19. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4, including durvalumab and tremelimumab if the following are fulfilled:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * All AEs of prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a ≥ Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE and not have experienced recurrence of an AE if re-challenged.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Nasopharyngeal carcinoma
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
4. >4 prior treatment lines with systemic therapy
5. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) ≤ 30 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator.
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
7. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg. hormone replacement therapy) is acceptable.
8. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
9. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
10. History of allogenic organ transplantation.
11. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
12. Uncontrolled undercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
13. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
14. History of leptomeningeal carcinomatosis
15. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab + tremelimumab combination therapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
21. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
22. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute toxicities of the treatment | 3 months
  The rate of Grade 3-5 combination TTC-related toxicities within 12 weeks from the start of SBRT treatments. The results will be tabulated to examine their frequency, organ systems affected, severity, and relationship to study treatment.
  Terminology Criteria for Adverse Events (CTCAE) V4.03 will be used for grading of AEs. Investigators will provide their assessment of causality as 1) unrelated, 2) unlikely, 3) possibly related, 4) probably, or 5) definitely related.
Progression Free Survival (PFS) | 6 months
  To evaluate whether the combination SBRT with Durvalumab and Tremelimumab will improve the progression-free survival of patients.
  Response will be assessed as per RECIST version 1.1.

SECONDARY OUTCOMES:
Local control (LC) | 2 years
  Defined as stable disease, partial response, or complete response based on serial imaging with CT scan. Recurrence will be defined as a suspicious mass at the site of SBRT treated lesion, progressing in size on 2 consecutive computed tomography scans at a minimum interval of 1 month, combined with a positive FDG-PET defined by a SUV max ≥ 5, or a biopsy-proven confirmation.
Progression-free survival (PFS) | 2 years
  Regional or distant disease progression according to RECIST v1.1 or death due to any cause
Overall survival (OS) | 2 years
  A subject will be classified as either alive or dead due to any cause. The time to event will be calculated as the time from Day 1 until date of death. Day 1 is the date of 1st treatment with durvalumab and tremelimumab.
Abscopal events | 2 years
  Defined as anti-tumor response outside the radiotherapy field.
  Response will be assessed as per RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

REFERENCES:
- [Derived] Bahig H, Aubin F, Stagg J, Gologan O, Ballivy O, Bissada E, Nguyen-Tan FP, Soulieres D, Guertin L, Filion E, Christopoulos A, Lambert L, Tehfe M, Ayad T, Charpentier D, Jamal R, Wong P. Phase I/II trial of Durvalumab plus Tremelimumab and stereotactic body radiotherapy for metastatic head and neck carcinoma. BMC Cancer. 2019 Jan 14;19(1):68. doi: 10.1186/s12885-019-5266-4. PMID 30642290